CLINICAL TRIAL: NCT00307190
Title: Postprandial Cholecystokinin Release and Gastric Emptying in Binge Eating Disorder
Brief Title: Hormone Release and Stomach Disturbances in People With Binge Eating Disorder
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #4735/#5797R; R01MH042206-04 (NIH); DATR A2-AID
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Binge Eating Disorder; Obesity; Eating Disorders
Keywords: BED
MeSH Terms: conditions — Binge-Eating Disorder; Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Binge Eating Disorder: Women with Binge Eating Disorder
- Controls: Weight, age, and gender-matched control subjects

SUMMARY:
This study will determine whether the disturbances in cholecystokinin release and gastric emptying that occur in people with binge eating disorder are similar to those that occur in people with bulimia nervosa.

DETAILED DESCRIPTION:
Binge Eating Disorder (BED) is a serious eating disorder that can occur in people of any weight, but occurs most frequently in people who are overweight. BED is characterized by the following eating behaviors: frequent episodes of eating large quantities of food in short periods of time; feeling out of control over one's eating behavior; feeling ashamed or disgusted by one's eating behavior; eating when not hungry; and eating in secret. BED is similar to Bulimia Nervosa (BN), in that binge eating is a characteristic of both disorders. However, people with BED do not purge after an episode of binge eating, and therefore often become overweight. The health risks of BED include those that are most commonly associated with clinical obesity. High blood pressure, high cholesterol levels, heart disease, diabetes mellitus, and gallbladder disease are all health problems that occur frequently in people with BED. CCK is a hormone that is released by the small intestine, and functions as a trigger for digestion and hunger suppression. People with BN often have disturbances in the release of cholecystokinin (CCK), which may contribute to their binge eating behavior. This study will determine whether the disturbances in CCK release and gastric emptying that occur in people with BED are similar to those that occur in people with BN.

Participants in this study will report to the study site on two non-consecutive days within a 2-week period for gastric emptying testing. On the day before the first study visit, participants will be instructed to eat a standardized dinner that does not include alcohol before 7 P.M., and not to eat or drink after 9 P.M. On the first day of testing, participants will lie in a semi-reclined position while drinking 600 ml of Ensure Plus. A gamma camera will be placed over the stomach to measure gastric emptying. In addition, a catheter will be inserted into the forearm of all participants for periodic blood testing throughout the process. On the second day of testing, participants will perform the same procedures, but the Ensure Plus will also contain a small amount of radioactive material so that gastric emptying can be tracked by the gamma camera. The testing procedure on each day will take approximately 90 minutes.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00308776

http://clinicaltrials.gov/show/NCT00304187

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Obese (body mass index (BMI) greater than 35 kg/m2)

For participants with BED:

* Meets DSM-IV criteria for BED
* BED duration of at least 1 year

For healthy participants:

* Weight close to that of participants with BED

Exclusion Criteria for all participants:

* Current or past diagnosis of BN, or any binge eating or self-induced vomiting
* Significant medical illness
* Current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder as defined by DSM-IV-TR
* Current DSM-IV-TR diagnosis of organic mental disorder, factitious disorder, or malingering
* History of a personality disorder (e.g., schizotypal, borderline, or antisocial) that might interfere with assessment or compliance with the study procedures
* At risk for suicide
* Currently taking psychotropic medication or medication that is known to affect appetite or gastric functioning
* History of drug or alcohol abuse within the 3 months prior to study entry
* Pregnant, planning to become pregnant, or lactating
* Anemia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, obese women between ages 18 and 60 with and without Binge Eating Disorder
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2004-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. T. Walsh, MD, Principal Investigator — New York State Psychiatric Institute at Columbia University Medical Center
Locations (1):
- Eating Disorders Clinic, New York State Psychiatric Institute, New York, New York, United States